CLINICAL TRIAL: NCT05238311
Title: Pre-approval Single-patient Expanded Access for Elranatamab (PF-06863135)
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C107; NCT05238311 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: refractory; relapsed
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Elranatamab

SUMMARY:
Provide pre-approval single-patient Expanded Access (Compassionate Use) of elranatamab for patients with relapsed/refractory multiple myeloma

DETAILED DESCRIPTION:
In Expanded Access, treating physicians are the Sponsors

Expanded Access requests from treating physicians should be directed to www.pfizercares.com Availability will depend on location.

ELIGIBILITY:
Must have relapsed/refractory multiple myeloma (RRMM) and be refractory to at least one immunomodulatory drug, one proteasome inhibitor and one anti-CD38 antibody. Must have evidence of disease progression after last therapy. Must have exhausted all available treatment options accessible as local standard of care and not be eligible for participation in any ongoing clinical trial. Additional eligibility criteria may be required.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult